CLINICAL TRIAL: NCT04612361
Title: Can Clinical Insomnia and Sleep Deprivation be a Cause of Adverse Maternal-fetal Outcome Among Egyptian Females in Their Last Trimester of Pregnancy;a Prospective Cohort Study
Brief Title: Effect of Clinical Insomnia and Sleep Deprivation on Maternal-fetal Outcome Among Egyptian Females in 3rd Trimester
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Dr. Osman Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Dr Hisham Gouda, Assistant Professor, Dr. Osman Hospital
Other Study IDs: Cairo University
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: Effect of Insomnia and Sleep Deprivation in 3rdtrimester
Keywords: insomnia,sleep deprivation,adverse maternal,fetal outcome
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non impaired sleep group: about 200-250 patients
  Interventions: Other: insommnia severity index questionnaire
- insomnia group: about 200 patients
  Interventions: Other: insommnia severity index questionnaire
- sleep deprived group: about 200-250 patients
  Interventions: Other: insommnia severity index questionnaire

INTERVENTIONS:
Other: insommnia severity index questionnaire — insomnia severity index questionnaire and scoring system

SUMMARY:
This prospective observational study aims at investigating whether insomnia or sleep deprivation during the 3rd trimester of pregnancy can be implicated in the occurrence of adverse maternal or fetal outcome. Data will be collected from all participants with special emphasis on: history of impaired sleep due to insomnia or sleep deprivation due to working on night shifts, history of insomnia during first 20 weeks of pregnancy.Number of night sleep hours and total number of sleep hours during the day will be recorded for each participant. The Insomnia severity index(ISI) a brief self report questionnaire used for assessing the degree of current insomnia will be administered to all participants at the time of their routine antenatal care visits to detect insomnia and its severity if present .The possible relationship between clinical insomnia or sleep deprivation and the occurrence of preterm birth or IUGR will be explored and the association with increased Cesarean delivery rate or painful and/ or prolonged labour.

DETAILED DESCRIPTION:
The demographic data will be collected from all participants including patient's age , BMI , gestational age, personal,present and past obstetric history, with special emphasis on: history of impaired sleep due to insomnia or sleep deprivation due to working on night shifts, history of insomnia during first 20 weeks of pregnancy.Number of night sleep hours and total number of sleep hours during the day will be recorded for each participant. The Insomnia severity index(ISI) a brief self report questionnaire used for assessing the degree of current insomnia will be administered to all participants at the time of their routine antenatal care visits to detect insomnia and its severity if present .It will be applied both in English and in its Arabic translated version. The ISI comprises seven items assessing the type of insomnia problem, satisfaction with the current sleep pattern, affection of the quality of life by the sleep problem, the degree of distress related to insomnia and its affect on daily functioning .Each item is scored on a scale of 0-4 and the total ISI score ranges from 0-28, with higher scores indicating more severe insomnia. A written informed consent will be obtained from each participant before joining the study. The participants will be followed up throughout their 3rd trimester till the time of their delivery. Any drop-out cases will be reported. The pregnant women who didn't suffer insomnia in any of the assessments, nor were sleep deprived due to working on night shifts will comprise the the non impaired sleep group and those suffering clinical insomnia as detected by the insomnia severity index (total score > or equal to 15) in any or all of the assessments will comprise the insomnia group. The 3rd group (sleep deprived group) will be comprised of participants who are only sleep deprived due to working on night shifts and not due to insomnia. Those getting less than 7hours of sleep/day will be considered sleep deprived.

The patients will be assessed during their routine visits with transabdominal ultrasound and Doppler studies for evaluation of fetal growth ,fetal well being ,placenta and exclusion of congenital anomalies, abnormal fetal position or presentation .The gestational age at delivery,mode of delivery,presence of prolonged or painful labour and fetal birth weight will all be recorded for comparison.

ELIGIBILITY:
Inclusion Criteria:The inclusion criteria will be ≥ 28 weeks gestational age as confirmed by first trimester scan or reliable 1st day of LMP ,normal singleton pregnancy , literate with no history of previous preterm birth or Cesarean delivery.

-

Exclusion Criteria Women with history of medical disorders with pregnancy, BMI≥ 30 , placenta previa, recent urinary tract or vaginal infections or obstetric complications during the current pregnancy or risk factors for preterm labour will be excluded. Women with history of diagnosed psychiatric disorder will be also excluded

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: * 28 weeks gestational age as confirmed by first trimester scan or reliable 1st day of LMP ,normal singleton pregnancy , literate with no history of previous preterm birth or Cesarean delivery. , with special emphasis on: history of impaired sleep due to insomnia or sleep deprivation due to working on night shifts, history of insomnia during first 20 weeks of pregnancy.Number of night sleep hours and total number of sleep hours during the day
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-10-30 (Estimated); Primary Completion 2021-03-28 (Estimated); Study Completion 2021-04-05 (Estimated)

PRIMARY OUTCOMES:
To explore possible relationship between clinical insomnia or sleep deprivation and the occurrence of preterm birth or IUGR | 6 months
  number of preterm deliveries and number of IUGR among the studied groups

SECONDARY OUTCOMES:
to evaluate whether insomnia or sleep deprivation are associated with increased Cesarean delivery rate or painful labour. | 6 months
  Number of cesarean deliveries among the 3 studied groups

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Hospitals,Obstetric clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided